CLINICAL TRIAL: NCT02182843
Title: Cellentra Viable Cell Bone Matrix (VCBM) Anterior Cervical Discectomy and Fusion Outcomes Study (VCBM/MaxAn)
Acronym: VCBM/ACDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-092
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Cervical Disc Degenerative Disorder
Keywords: Cellentra ACDF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cellentra VCBM (Experimental): Cellentra™ VCBM is an allogenic bone graft containing naturally occurring viable donor cells intended for homologous use in the repair, replacement, reconstruction or supplementation of the recipient's tissue in musculoskeletal defects.
  Interventions: Biological: Cellentra VCBM

INTERVENTIONS:
Biological: Cellentra VCBM — Cellentra™ VCBM is an allogenic bone graft containing naturally occurring viable donor cells intended for homologous use in the repair, replacement, reconstruction or supplementation of the recipient's tissue in musculoskeletal defects.

SUMMARY:
The purpose of this study is to assess the clinical and radiographic outcomes in patients who undergo ACDF procedures using Cellentra Viable Cell Bone Matrix (VCBM), cortical allograft spacers, and the MaxAn® Anterior Cervical Plate System. Cellentra VCBM will be compared to published data for autograft in NDI (Neck Disability Index) improvement and radiographic success of fusion.

DETAILED DESCRIPTION:
This is a prospective single-arm multi-center study of Cellentra Viable Cell Bone Matrix (VCBM) and the MaxAn® Anterior Cervical Plate System when used in anterior cervical discectomy and fusion procedures. This study will enroll up to eighty (80) subjects across up to eight (8) clinical sites. Subjects will be recruited from a pool of patients presenting to investigators for an anterior cervical discectomy and fusion procedure.

ELIGIBILITY:
Inclusion Criteria:

* The subject is scheduled to undergo a two or three level primary spinal fusion surgery between the levels of C2-T1 (Cervical 2 to Thoracic 1) using Cellentra™ VCBM, allograft spacers, and the MaxAn® Anterior Cervical Plate System.
* The subject is 18 years of age or older.
* The subject was unresponsive to conservative treatment for at least 6 weeks unless clinically indicated sooner.
* The subject has persistent neck, shoulder, or arm pain consistent with cervical degenerative disc disease confirmed by patient history and radiographic studies.
* The subject must in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent.

Exclusion Criteria:

1. Subject has an active local or systemic infection.
2. Subject is morbidly obese, defined as a BMI greater than 40.
3. Subject has a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the investigator's opinion may interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up.
4. Subject has inadequate tissue coverage over the operative site.
5. Subject has an open wound local to the operative area, or rapid joint disease, bone absorption, osteopenia, osteomalacia and/or osteoporosis.
6. Any previous cervical spinal surgery.
7. Subject has a condition requiring medications that may interfere with bone or soft tissue healing (i.e., oral or parenteral glucocorticoids, immunosuppressives, methotrexate, etc.) or immunocompromised.
8. Subject has any medical condition or extenuating circumstance that, in the opinion of the investigator, would preclude participation in the study.
9. Subject who does not meet the specific indications for use of the Cellentra™ VCBM or MaxAn® Anterior Cervical Plate System.
10. Subject is pregnant, lactating or interested in becoming pregnant during the duration of the study.
11. Subject is currently involved in another investigational drug or device study that could confound study data.
12. Subject is a prisoner.
13. Subject has a metal sensitivity/foreign body sensitivity.
14. Subject is involved in or planning to engage in litigation or receiving Worker's Compensation related to neck or back pain.
15. Subject has sensitivity or allergies to any of the processing agents. (See package insert for Cellentra™ VCBM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Batts, Study Director — Biomet Spine
Locations (6):
- United States (6):
  - Barrow Neurological Associates, Phoenix, Arizona
  - Fort Wayne Ortho, Fort Wayne, Indiana
  - Orthopaedic Institute of Western KY, Paducah, Kentucky
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Rothman Institute, Philadelphia, Pennsylvania
  - Spine Team Texas, Southlake, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gore DR, Sepic SB. Anterior cervical fusion for degenerated or protruded discs. A review of one hundred forty-six patients. Spine (Phila Pa 1976). 1984 Oct;9(7):667-71. doi: 10.1097/00007632-198410000-00002. PMID 6505833
- [Background] Palit M, Schofferman J, Goldthwaite N, Reynolds J, Kerner M, Keaney D, Lawrence-Miyasaki L. Anterior discectomy and fusion for the management of neck pain. Spine (Phila Pa 1976). 1999 Nov 1;24(21):2224-8. doi: 10.1097/00007632-199911010-00009. PMID 10562988
- [Background] McConnell JR, Freeman BJ, Debnath UK, Grevitt MP, Prince HG, Webb JK. A prospective randomized comparison of coralline hydroxyapatite with autograft in cervical interbody fusion. Spine (Phila Pa 1976). 2003 Feb 15;28(4):317-23. doi: 10.1097/01.BRS.0000048503.51956.E1. PMID 12590203
- [Background] Samartzis D, Shen FH, Goldberg EJ, An HS. Is autograft the gold standard in achieving radiographic fusion in one-level anterior cervical discectomy and fusion with rigid anterior plate fixation? Spine (Phila Pa 1976). 2005 Aug 1;30(15):1756-61. doi: 10.1097/01.brs.0000172148.86756.ce. PMID 16094278
- [Background] Bridwell KH, Lenke LG, McEnery KW, Baldus C, Blanke K. Anterior fresh frozen structural allografts in the thoracic and lumbar spine. Do they work if combined with posterior fusion and instrumentation in adult patients with kyphosis or anterior column defects? Spine (Phila Pa 1976). 1995 Jun 15;20(12):1410-8. PMID 7676341
- [Background] Soderlund CH, Pointillart V, Pedram M, Andrault G, Vital JM. Radiolucent cage for cervical vertebral reconstruction: a prospective study of 17 cases with 2-year minimum follow-up. Eur Spine J. 2004 Dec;13(8):685-90. doi: 10.1007/s00586-004-0747-8. Epub 2004 Jun 26. PMID 15662542
- [Background] Fountas KN, Kapsalaki EZ, Nikolakakos LG, Smisson HF, Johnston KW, Grigorian AA, Lee GP, Robinson JS Jr. Anterior cervical discectomy and fusion associated complications. Spine (Phila Pa 1976). 2007 Oct 1;32(21):2310-7. doi: 10.1097/BRS.0b013e318154c57e. PMID 17906571
- [Background] Carreon LY, Glassman SD, Campbell MJ, Anderson PA. Neck Disability Index, short form-36 physical component summary, and pain scales for neck and arm pain: the minimum clinically important difference and substantial clinical benefit after cervical spine fusion. Spine J. 2010 Jun;10(6):469-74. doi: 10.1016/j.spinee.2010.02.007. Epub 2010 Apr 1. PMID 20359958
- [Background] Young BA, Walker MJ, Strunce JB, Boyles RE, Whitman JM, Childs JD. Responsiveness of the Neck Disability Index in patients with mechanical neck disorders. Spine J. 2009 Oct;9(10):802-8. doi: 10.1016/j.spinee.2009.06.002. Epub 2009 Jul 25. PMID 19632904
- [Background] Coric D, Nunley PD, Guyer RD, Musante D, Carmody CN, Gordon CR, Lauryssen C, Ohnmeiss DD, Boltes MO. Prospective, randomized, multicenter study of cervical arthroplasty: 269 patients from the Kineflex|C artificial disc investigational device exemption study with a minimum 2-year follow-up: clinical article. J Neurosurg Spine. 2011 Oct;15(4):348-58. doi: 10.3171/2011.5.SPINE10769. Epub 2011 Jun 24. PMID 21699471
- [Background] Davis RJ, Kim KD, Hisey MS, Hoffman GA, Bae HW, Gaede SE, Rashbaum RF, Nunley PD, Peterson DL, Stokes JK. Cervical total disc replacement with the Mobi-C cervical artificial disc compared with anterior discectomy and fusion for treatment of 2-level symptomatic degenerative disc disease: a prospective, randomized, controlled multicenter clinical trial: clinical article. J Neurosurg Spine. 2013 Nov;19(5):532-45. doi: 10.3171/2013.6.SPINE12527. Epub 2013 Sep 6. PMID 24010901
- [Background] Lofgren H, Engquist M, Hoffmann P, Sigstedt B, Vavruch L. Clinical and radiological evaluation of Trabecular Metal and the Smith-Robinson technique in anterior cervical fusion for degenerative disease: a prospective, randomized, controlled study with 2-year follow-up. Eur Spine J. 2010 Mar;19(3):464-73. doi: 10.1007/s00586-009-1161-z. Epub 2009 Sep 18. PMID 19763634
- [Background] Miller LE, Block JE. Safety and effectiveness of bone allografts in anterior cervical discectomy and fusion surgery. Spine (Phila Pa 1976). 2011 Nov 15;36(24):2045-50. doi: 10.1097/BRS.0b013e3181ff37eb. PMID 21304437
- [Background] Mummaneni PV, Burkus JK, Haid RW, Traynelis VC, Zdeblick TA. Clinical and radiographic analysis of cervical disc arthroplasty compared with allograft fusion: a randomized controlled clinical trial. J Neurosurg Spine. 2007 Mar;6(3):198-209. doi: 10.3171/spi.2007.6.3.198. PMID 17355018

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cellentra VCBM
Started | 81
Completed | 71
Not Completed | 10
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cellentra VCBM
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 72
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 81
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (5.4)
Tobacco Use [Count of Participants; unit: Participants]
  Current | 31
  Past | 12
  Never | 38
Previous Spine Surgery [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in NDI From Baseline
Description: Neck Disability Index (NDI) is a patient-completed, condition-specific functional status questionnaire including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Each of the 10 items is scored from 0 - 5, with a maximum score of 50. The obtained score is multiplied by 2 to produce a percentage score. A higher score indicates more patient-rated disability (0 points or 0% means : no activity limitations , 50 points or 100% means complete activity limitation). The minimal clinically important difference or change (MCID / MCIC) is described as the smallest difference or change that patients perceive as beneficial. In patients with cervical radiculopathy the MCID is 7 points of change ( 14%). In order to demonstrate improvement in status, the NDI would need to be reduced by at least 14%.
Time Frame: 12 months after device implantation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cellentra VCBM
Number analyzed (Participants) | 81
score on a scale
  Baseline | 52.1 (19.1)
  12 months | 28.5 (24.3)
  Mean Change in NDI | 24.0 (21.9)

2. Secondary Outcome: Number of Participants With Radiographic Success at 24 Months
Description: Radiographic fusion was assessed at each operated level using the Bridwell fusion grading system:
  * Grade I (definite) - Fused with remodeling and trabeculae
  * Grade II (probable) - Graft intact, not fully remodeled and incorporated through, no lucencies
  * Grade III (probably not) - Graft intact, but definite lucency at the top or bottom of the graft
  * Grade IV (no) - Definitely not fused, with resorption of bone graft or collapse.
  Radiographic success was defined as grade 1 or 2 fusion at every operated level at 24 months
Time Frame: 24 Months
Population: 71/81 of originally enrolled participants had radiographs available for analysis at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cellentra VCBM
Number analyzed (Participants) | 71
Participants | 35

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of surgery through last follow up at 24 months.
Description: All clinical events, including both observed or volunteered problems, complaints, symptoms, physical signs or disease which either occur during the study, having been absent at baseline, or, if present at baseline, appear to worsen during the clinical outcomes collection study are to be recorded as complications in the subject's medical record and on the appropriate case report form.
Arm/Group | Cellentra VCBM
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 8/81
Other Adverse Events (participants affected / at risk) | 43/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cellentra VCBM (N=81)
Lumbar Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Cerbrovascular ischemia (Nervous system disorders) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cellentra VCBM (N=81)
Autoimmune disorder (Immune system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cerebrospinal fluid leak (Nervous system disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Delayed union (Musculoskeletal and connective tissue disorders) | 7 (7)
Dural defect (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 6 (6)
Headache (Nervous system disorders) | 2 (2)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain (General disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Radiculitis (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT02182843/Prot_SAP_000.pdf